CLINICAL TRIAL: NCT04356690
Title: A Phase II Single-Center, Randomized, Open-Label, Safety and Efficacy Study of Etoposide in Patients With COVID-19 Infection
Brief Title: Etoposide in Patients With COVID-19 Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual, change in COVID prevalence, availability of effective vaccine
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, John Mark Sloan, Principal Investigator, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-40102
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: Etoposide; hemophagocytic lymphohistiocytosis (HLH); cytokine storm
MeSH Terms: conditions — COVID-19; Lymphohistiocytosis, Hemophagocytic; Cytokine Release Syndrome | interventions — Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 - Etoposide (Experimental): Participants that are on ventilation Etoposide 150 mg/m2 daily days 1 and 4
  Interventions: Drug: Etoposide
- Cohort 1 - Control (No Intervention): Standard of care therapy in participants that are on ventilation

INTERVENTIONS:
Drug: Etoposide — Etoposide 150 mg/m2 administered intravenously once daily on Days 1 and 4.
  Other Names: Etopophos
  Arms: Cohort 1 - Etoposide

SUMMARY:
This is a randomized, open-label phase II study designed to evaluate the safety and efficacy of etoposide in patients with the 2019 novel coronavirus (COVID-19) infection. Randomization will be performed with a 3:1 allocation ratio. Treatment will be comprised of etoposide administered intravenously at a dose of 150 mg/m2 on Days 1 and 4 in patients with COVID-19 infection meeting eligibility criteria. Subsequent doses of etoposide will be allowed if the investigator and treating physician believe the patient had clinical benefit from etoposide therapy but subsequently has evidence of recurrent clinical deterioration. Subjects randomized to control will receive standard of care treatment. No placebo will be used.

DETAILED DESCRIPTION:
The rationale for the use of etoposide to treat the cytokine storm in COVID-19 is the high mortality associated with the hyperinflammatory response to the virus, which is similar to that seen in other secondary types of Hemophagocytic lymphohistiocytosis. Autopsy studies of Acute respiratory distress syndrome (ARDS) in COVID patients show a high number of cytolytic T cells in the lungs of such patients. Early autopsy results of COVID patients at Boston Medical Center demonstrate significant hemophagocytosis in lymph nodes and spleen. Comparable studies in the related coronavirus infection severe acute respiratory syndrome (SARS) have demonstrated hemophagocytosis, a hallmark of HLH.15 By targeting the T cells and monocytes driving the cytokine storm in patients with the more severe forms of COVID infection, we hope to alleviate the progression of lung and multi-organ dysfunction characteristic of patients who die from this illness.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 infection
* Evidence of cytokine storm defined as:

  * Peak ferritin > 10,000 ng/mL OR
  * Peak ferritin > 500 ng/mL and one or more of the following at any time during hospital admission: Lactate dehydrogenase > 500 U/L, d-dimer >1000 ng/mL, C-reactive protein > 100 mg/L, or white blood count> 15 k/microlitre

Cohort 1: Intubated status as a result of COVID infection-associated respiratory illness.

Exclusion Criteria:

* Pregnancy or breastfeeding
* History of severe hypersensitivity to etoposide products
* Absolute neutrophil count (ANC) < 1000 cells/mm3
* Platelet count <50,000/mm3
* Bilirubin > 3.0 mg/dL
* Aspartate OR alanine aminotransferase > 5.0 x upper limit of normal
* Creatinine Clearance < 15 mL/min (calculated by Cockcroft Fault formula)
* Requiring continuous renal replacement therapy
* Requiring >1 vasopressor
* Requiring extracorporeal membrane oxygenation (ECMO)
* Other active, life-threatening infections
* Anti-cytokine treatment (including anakinra or Interleukin 6 antibodies eg tocilizumab, sarilumab) administration within three half-lives of the medication used
* Hydroxychloroquine, colchicine, azithromycin, doxycycline-if administered for COVID infection-must be discontinued for at least 24 hours prior to randomization.
* Has a history or current evidence of any condition, therapy or laboratory abnormality that might confound the results of the study, interfere with subject participation, or is not in the best interest of the patient to participate, in the opinion of the investigator.
* Inability to consent and no legally authorized representative
* Poorly controlled HIV infection (CD4 count <100 cells/mm3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mark Sloan, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 - Etoposide | Cohort 1 - Control
Started | 6 | 2
Completed | 6 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Etoposide | Cohort 1 - Control | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Continuous [Median (Full Range); unit: years] | 62.5 [51 to 87] | 74.5 [71 to 78] | 67 [51 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black or African American | 1 | 0 | 1
  White | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8
Baseline Ferritin Blood Levels [Mean (Standard Deviation); unit: ng/ml] | 1754.17 (797.34) | 2699.5 (3270.37) | 1990.5 (1474.28)
Baseline white blood cell counts [Mean (Standard Deviation); unit: cells x1000 per mL] | 12.57 (7.79) | 16.75 (4.45) | 13.61 (7.07)
Baseline C Reactive protein levels [Mean (Standard Deviation); unit: mg/L] | 151.17 (130.15) | 145.50 (111.02) | 149.75 (117.76)
Baseline d-dimer blood levels [Mean (Standard Deviation); unit: ng/ml DDU] | 1394.00 (1183.31) | 4745.00 (6167.39) | 2231.75 (2973.25)
Baseline platelet counts [Mean (Standard Deviation); unit: cells x 1000 per mL] | 274.50 (193.45) | 274.50 (126.57) | 274.50 (170.35)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Pulmonary Status by Two Categories on an 8 Point Ordinal Scale of Respiratory Function
Description: 8-Point Ordinal Scale of Respiratory Function: 8 -Death; 7 -Ventilation in addition to extracorporeal membrane oxygen (ECMO), continuous renal replacement therapy (CRRT), or need for vasopressors (dopamine ≥5 μg/kg/min OR epinephrine ≥0.1 μg/kg/min OR norepinephrine ≥0.1 μg/kg/min) 6 -Intubation and mechanical ventilation 5 -Non-invasive mechanical ventilation (NIV) or high-flow oxygen 4 -Hospitalized, requiring oxygen by mask or nasal prongs 3 -Hospitalization without oxygen supplementation 2-Discharged from hospital either to home with supplemental oxygen OR to inpatient rehabilitation/skilled nursing facility(+/-supplemental oxygen);
  1 -Discharged to home without supplemental oxygen
Time Frame: baseline, through hospital discharge or death
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Etoposide | Cohort 1 - Control
Number analyzed (Participants) | 6 | 2
Participants | 2 | 1

2. Secondary Outcome: Overall Survival
Description: Number of participants that lived to day 30 or hospital discharge
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Etoposide | Cohort 1 - Control
Number analyzed (Participants) | 6 | 2
Participants | 3 | 1

3. Secondary Outcome: Length of Hospitalization
Description: Number of days participants were hospitalized after treatment
Time Frame: From date of enrollment until date of discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1 - Etoposide | Cohort 1 - Control
Number analyzed (Participants) | 6 | 2
days | 17 (11.35) | 24 (5.66)

4. Secondary Outcome: Duration of Ventilation After Treatment
Description: Number of days participants were ventilated after treatment
Time Frame: From date of enrollment until the date of extubation
Population: 4 participants who were not extubated before death are excluded- 3 in Etoposide arm and 1 in the Control arm.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1 - Etoposide | Cohort 1 - Control
Number analyzed (Participants) | 3 | 1
days | 15.67 (12.9) | 15.0 (0)

5. Secondary Outcome: Change in Blood Ferritin Levels
Description: Change in ferritin from treatment to day 30
Time Frame: baseline, to day 30 (or discharge or death)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 - Etoposide | Cohort 1 - Control
Number analyzed (Participants) | 6 | 2
ng/mL | 1235.67 (1180.59) | -1771.50 (2320.02)

6. Secondary Outcome: Change in C-reactive Protein (CRP) Levels
Description: Change in CRP levels from treatment to day 30
Time Frame: baseline, to day 30 (or discharge or death)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cohort 1 - Etoposide | Cohort 1 - Control
Number analyzed (Participants) | 6 | 2
mg/L | -49.00 (64.38) | -74.00 (63.64)

7. Secondary Outcome: Change in D-dimer Blood Levels
Description: Change in d-dimer from treatment to day 30
Time Frame: baseline, to day 30 (or discharge or death)
Measure: Mean (Standard Deviation); unit: mg/ml DDU
Arm/Group | Cohort 1 - Etoposide | Cohort 1 - Control
Number analyzed (Participants) | 6 | 2
mg/ml DDU | 480.67 (2427.12) | -2243.00 (3618.97)

8. Secondary Outcome: Change in White Blood Cell Count
Description: Change in white blood cell count from treatment to day 30
Time Frame: baseline, to day 30 (or discharge or death)
Measure: Mean (Standard Deviation); unit: cells x 1000 per mL
Arm/Group | Cohort 1 - Etoposide | Cohort 1 - Control
Number analyzed (Participants) | 6 | 2
cells x 1000 per mL | 5.18 (6.35) | 13.40 (10.04)

9. Secondary Outcome: Change in Platelet Count
Description: Change in platelet count from treatment to day 30
Time Frame: baseline, to day 30 (or discharge or death)
Measure: Mean (Standard Deviation); unit: cells x 1000 per mL
Arm/Group | Cohort 1 - Etoposide | Cohort 1 - Control
Number analyzed (Participants) | 6 | 2
cells x 1000 per mL | -70.00 (100.84) | 102.00 (72.12)

ADVERSE EVENTS:
Time Frame: Treatment/enrollment until discharge or death
Arm/Group | Cohort 1 - Etoposide | Cohort 1 - Control
All-Cause Mortality (participants affected / at risk) | 3/6 | 1/2
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/2
Other Adverse Events (participants affected / at risk) | 6/6 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Etoposide (N=6) | Cohort 1 - Control (N=2)
febrile neutropenia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Etoposide (N=6) | Cohort 1 - Control (N=2)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Thrombocytopenia
anemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) — anemia
neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) — neutropenia
Abnormal LFTs (Hepatobiliary disorders) | 1 (1) | 0 (0) — Abnormal LFTs
acute kidney innury (Renal and urinary disorders) | 1 (1) | 1 (1) — acute kidney injury
ventilatory asscociated pneumonia (Infections and infestations) | 1 (1) | 0 (0) — ventilator associated pneumonia (non-neutropenic)

LIMITATIONS AND CAVEATS:
The study was halted prematurely due to slow accrual, change in COVID prevalence, and the availability of an effective vaccine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT04356690/Prot_SAP_000.pdf